CLINICAL TRIAL: NCT02695498
Title: Mindfulness and Mechanisms of Pain Processing in Adults With Migraines
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB00027845-B; K23AT008406 (NIH)
Record Dates: First submitted 2016-01-11; First posted 2016-03-01 (Estimated); Results first posted 2023-11-27 (Actual); Last update posted 2023-11-27 (Actual); Status verified 2019-08

CONDITIONS: Migraine
Keywords: migraine with aura; migraine without aura; pain; controls; mind-body
MeSH Terms: conditions — Migraine Disorders; Migraine with Aura; Migraine without Aura; Pain | interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness Based Stress Reduction (Experimental): Mindfulness Based Stress Reduction (MBSR) is a standardized course in mindfulness mediation and yoga.
  Interventions: Other: Mindfulness Based Stress Reduction
- Migraine/stress Education (Experimental): This course will educate participants about migraine pathophysiology, headache triggers, stress, gentle stretches, and daily migraine readings.
  Interventions: Other: Migraine/stress Education

INTERVENTIONS:
Other: Mindfulness Based Stress Reduction — MBSR is a standardized course in mindfulness mediation and yoga. The participants will meet weekly for 8 weeks for 2.5 hours, plus a "mindfulness retreat day" (approximately 6 hours) after the 6th class [9 total classes.] Mindfulness is cultivated through meditation, body scan (sequential attention to parts of the body), and mindful movement (bodily awareness during gentle stretching, based on yoga). The instructor also gives information about stress and stress relief.
  Arms: Mindfulness Based Stress Reduction
Other: Migraine/stress Education — The participants will be educated about migraine pathophysiology, headache triggers, stress, gentle stretches, and daily migraine readings.
  Arms: Migraine/stress Education

SUMMARY:
Although many adults with migraines use non-pharmacological treatment options, there is a lack of research on the use of many mind/body techniques specifically for headache. This research will further the understanding of the mechanisms, efficacy, and predictors of mind-body practices in adults with migraines.

DETAILED DESCRIPTION:
Migraine is a common and disabling pain condition. Affective/cognitive processes, such as pain catastrophizing and emotional reactivity, often play a major role in migraine pain and disability. These processes may be just as important to target as the sensory aspect given their impact on outcomes and disability. Because of this cognitive/affective load that builds over time in migraine, we hypothesize A) migraineurs perceive affective pain processing differently than non-migraineurs and B) mind/body therapies that target these factors may be especially beneficial and may differentially impact the affective component of migraine pain. Evidence shows that meditation decreases affective (e.g., pain unpleasantness) over sensory (e.g., pain intensity) response to experimental pain and reduces pain by engaging brain regions important for cognitive and affective modulation of pain. By measuring both experimental and clinical pain, the study team will be able to test these hypotheses.

ELIGIBILITY:
Inclusion Criteria:

Diagnosis of migraine; ≥18yo; ≥1 yr of migraines; 4-20 days/month with migraines; able and willing to participate in 8 weekly sessions and daily homework 30-45min

Exclusion Criteria:

Current regular (weekly or more often) practice of meditation; any major unstable medical/psychiatric illness (e.g., hospitalization within 90 days, suicide risk, etc.); other non-migraine chronic pain condition (e.g., fibromyalgia, low back pain, etc.) or sensory abnormalities (e.g., neuropathy, Raynaud's, etc.); diagnosis of medication overuse headache; volunteers with no pain ratings to frankly noxious stimuli (temperatures > 49°C) or excessive responses to threshold temperatures (~43°C); current or planned pregnancy or breastfeeding, any new medication started within 4 weeks of screening visit; unwilling to maintain stable current medication dosages for duration of trial; failure to complete baseline headache logs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2016-08-26 (Actual); Primary Completion 2019-07-17 (Actual); Study Completion 2019-07-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca E Wells, MD, MPH, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Findings will be disseminated so that providers can implement the results into clinical practice, for scientists to build upon in their research, and for patients to inform treatment decisions. Results will be made publicly available through this website. In addition, results will be published in respected peer-reviewed journals, presented to colleagues at scientific meetings, and discussed with the press.
Supporting Information: Study Protocol
Access Criteria: Please contact Dr. Rebecca Wells for information regarding the study protocol and Institutional Review Board (IRB) approvals.

REFERENCES:
- [Background] Wells RE, Burch R, Paulsen RH, Wayne PM, Houle TT, Loder E. Meditation for migraines: a pilot randomized controlled trial. Headache. 2014 Oct;54(9):1484-95. doi: 10.1111/head.12420. Epub 2014 Jul 18. PMID 25041058
- [Derived] Wells RE, O'Connell N, Pierce CR, Estave P, Penzien DB, Loder E, Zeidan F, Houle TT. Effectiveness of Mindfulness Meditation vs Headache Education for Adults With Migraine: A Randomized Clinical Trial. JAMA Intern Med. 2021 Mar 1;181(3):317-328. doi: 10.1001/jamainternmed.2020.7090. PMID 33315046

RESULTS

PARTICIPANT FLOW:
Groups:
- Mindfulness Based Stress Reduction: Mindfulness Based Stress Reduction (MBSR) is a standardized course in mindfulness mediation and yoga.
  Mindfulness Based Stress Reduction: MBSR is a standardized course in mindfulness mediation and yoga.
  The participants will meet weekly for 8 weeks for 2.5 hours, plus a "mindfulness retreat day" (approximately 6 hours) after the 6th class [9 total classes.] Mindfulness is cultivated through meditation, body scan (sequential attention to parts of the body), and mindful movement (bodily awareness during gentle stretching, based on yoga). The instructor also gives information about stress and stress relief.
Period: Overall Study
Arm/Group | Mindfulness Based Stress Reduction | Migraine/Stress Education
Started | 45 | 44
Completed | 45 | 44
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mindfulness Based Stress Reduction | Migraine/Stress Education | Total
Number analyzed (Participants) | 45 | 44 | 89
Age, Continuous [Mean (Standard Deviation); unit: years] | 44 (12) | 44 (14) | 44 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 40 | 82
  Male | 3 | 4 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 4 | 6
  Not Hispanic or Latino | 43 | 40 | 83
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 5 | 10
  White | 40 | 39 | 79
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 45 | 44 | 89
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 27 (8) | 29 (7) | 28 (7.48)
Systolic Blood Pressure [Mean (Standard Deviation); unit: mm Hg] | 120 (16.5) | 122 (12.9) | 121 (14.6)
Diastolic Blood Pressure [Mean (Standard Deviation); unit: mm Hg] | 73 (11.4) | 73 (8.8) | 73 (10)
Heart Rate [Mean (Standard Deviation); unit: beats per minute] | 73 (13) | 78 (13) | 75.5 (13.4)

OUTCOME MEASURES:

1. Primary Outcome: Change in Frequency of Migraine Days Per Month From Baseline
Description: Change in frequency of migraine days from baseline: A migraine day is defined as a calendar day (00:00 to 23:59) when the patient reports 4 or more continuous hours of a moderate to severe headache (rating of 6-10 on 0-10 pain intensity scale) and/or they treated a headache with abortive medication; tracked with headache logs.
Time Frame: Baseline and immediately post-intervention (12 weeks)
Measure: Mean (95% Confidence Interval); unit: number of days
Arm/Group | Mindfulness Based Stress Reduction | Migraine/Stress Education
Number analyzed (Participants) | 45 | 44
number of days | -1.6 [-2.5 to -0.7] | -2.0 [-2.9 to -1.1]

2. Secondary Outcome: Change in Frequency of Migraine Days From Baseline
Description: as for outcome 1
Time Frame: 3 months post-intervention
Measure: Mean (95% Confidence Interval); unit: days
Arm/Group | Mindfulness Based Stress Reduction | Migraine/Stress Education
Number analyzed (Participants) | 45 | 44
days | -2.2 [-3.2 to -1.1] | -1.98 [-3.1 to -0.9]

3. Secondary Outcome: Change in Frequency of Headache Days From Baseline
Description: Change in frequency of any day with a headache tracked with headache logs
Time Frame: Baseline to Immediately post-intervention (12 weeks)
Population: only reporting 'headache' duration (not 'migraine' duration) (e.g., data were not collected)
Arm/Group | Mindfulness Based Stress Reduction | Migraine/Stress Education
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Change in Headache Duration From Baseline to 12 Weeks
Description: Modeled change in headache duration from baseline 4 weeks to weeks 8-12 by calculating the duration (in hours) of each headache attack and using a multivariable linear mixed model framework controlling for baseline value of the outcome of interest, treatment group, cohort, and within participant variation via random effects, with significance based on the treatment group effect and phase interaction at .05 significance level.
Time Frame: From baseline to Immediately post-intervention (12 weeks)
Population: Data were not collected)
Arm/Group | Mindfulness Based Stress Reduction | Migraine/Stress Education
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Change in Migraine Severity-pain Intensity From Baseline to Week 12
Description: change in headache severity-pain intensity from baseline 4 weeks to weeks 8-12. For each headache attack, participants rated the pain intensity on a 0-10 scale (0, no pain sensation, 10 most intense pain sensation imaginable). We calculated the pain intensity of each headache attack and used a multivariable linear model framework controlling for baseline value of the outcome of interest, treatment group, cohort, and within participant variation via random effects, with significance based on the treatment group effect and phase interaction at .05 significance level.
Time Frame: baseline to Week 12
Population: Our multivariable linear model resulted in a 95% confidence interval for the difference between the 2 values from the two Groups
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Mindfulness Based Stress Reduction | Migraine/Stress Education
Number analyzed (Participants) | 45 | 44
score on a scale | -0.142 [-0.738 to 0.0997] | -.177 [-0.738 to 0.0997]

6. Secondary Outcome: Change in Headache Severity-pain Intensity From Baseline to Week 12
Description: Modeled change in headache severity-pain intensity from baseline 4 weeks to weeks 8-12. For each headache attack, participants rated the pain intensity on a 0-10 scale (0, no pain sensation, 10 most intense pain sensation imaginable). Higher scores mean a worse outcome in terms of pain intensity.
Time Frame: Baseline and 12 weeks
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Mindfulness Based Stress Reduction | Migraine/Stress Education
Number analyzed (Participants) | 45 | 44
score on a scale | 0.142 [-0.156 to 0.440] | -0.177 [-0.472 to 0.117]

7. Secondary Outcome: Change in Migraine Severity-pain Unpleasantness From Baseline
Description: Change in migraine severity on 0-10 scale in pain unpleasantness from baseline (tracked with headache logs)
Time Frame: Baseline to 6 months post-intervention
Reporting Status: Not Posted

8. Secondary Outcome: Change in Headache Severity-pain Unpleasantness From Baseline to 12 Weeks
Description: Change in headache severity on 0-10 scale (0, "not at all unpleasant" to 10, "most unpleasant imaginable") in pain unpleasantness from baseline 4 weeks to weeks 8-12 (tracked with headache logs).
Time Frame: Baseline and 12 weeks
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Mindfulness Based Stress Reduction | Migraine/Stress Education
Number analyzed (Participants) | 45 | 44
score on a scale | .1745 [-0.189 to 0.538] | -0.0884 [-0.447 to 0.270]

9. Secondary Outcome: Percent Change in Score in Response to Experimental Heat Pain on Pain Intensity Measure From Baseline (0-10) Visual Analogue Scale (VAS Scale ) to 12 Weeks
Description: Using a 10 cm sliding visual analogue scale, participants quantified intensity (from "no pain sensation" to "most intense imaginable"), at baseline and at 12 weeks for each of 6 measures at 49 °C. A multivariable linear mixed model was used to model the percent change from baseline in perceived pain intensity at each visit for each of 6 measures at 49 °C. The VAS consists of a 10cm line, with two end points representing 0 ('no pain') and 10 ('pain as bad as it could possibly be'). Ask the patient to rate their current level of pain by placing a mark on the line.
Time Frame: Baseline to week 12
Measure: Mean (95% Confidence Interval); unit: percentage of change
Arm/Group | Mindfulness Based Stress Reduction | Migraine/Stress Education
Number analyzed (Participants) | 45 | 44
percentage of change | -36.3 [-60.3 to -12.3] | 13.5 [-9.9 to 36.8]

10. Secondary Outcome: Percent Change in Response Score to Experimental Heat Pain on Pain Unpleasantness Measure From Baseline (0-10) Visual Analogue Scale (VAS Scale) From Baseline to 12 Weeks
Description: Using a 10 cm sliding visual analogue scale, participants quantified unpleasantness (from "not at all unpleasant" to "most unpleasant imaginable"). Participants rated perceived pain unpleasantness at baseline and at 12 weeks for each of 6 measures at 49 °C. A multivariable linear mixed model was used to model the percent change from baseline in perceived pain intensity at each visit for each of 6 measures at 49 °C. Change scores were modeled as a function of treatment group and visit, controlling for baseline. The VAS consists of a 10cm line, with two end points representing 0 ('no pain') and 10 ('pain as bad as it could possibly be'). Ask the patient to rate their current level of pain by placing a mark on the line.
Time Frame: Baseline to week 12
Measure: Mean (95% Confidence Interval); unit: percentage of change
Arm/Group | Mindfulness Based Stress Reduction | Migraine/Stress Education
Number analyzed (Participants) | 45 | 44
percentage of change | -30.4 [-49.4 to -9.9] | 11.2 [-8.9 to 31.2]

11. Secondary Outcome: Change in Experimental Heat Pain Threshold From Baseline to Week 12
Description: Change in Experimental Heat Pain Threshold From Baseline to 12 weeks
Time Frame: Baseline to week 12
Measure: Mean (95% Confidence Interval); unit: Degree Celsius
Arm/Group | Mindfulness Based Stress Reduction | Migraine/Stress Education
Number analyzed (Participants) | 45 | 44
Degree Celsius | 0.096 [-0.656 to 0.858] | 0.162 [-0.619 to 0.943]

12. Secondary Outcome: Change in Headache-related Disability From Baseline
Description: Change in headache-related disability from baseline (Migraine Disability Assessment (MIDAS)-one month) Score range is 0-21+
  0 to 5: MIDAS grade I, little or no disability 6 to 10: MIDAS grade II, mild disability 11 to 20: MIDAS grade III, moderate disability 21 or higher: MIDAS grade IV, severe disability
Time Frame: Baseline to Immediately post-intervention
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Mindfulness Based Stress Reduction | Migraine/Stress Education
Number analyzed (Participants) | 45 | 44
score on a scale | -7.6 [-10.1 to -5.0] | -1.7 [-4.1 to 0.8]

13. Secondary Outcome: Change in Headache Disability Scores From Baseline
Description: Change in headache-related disability from baseline ( Headache Impact Test (HIT)-6)
  Headache impact severity level can be categorized using score ranges based on the HIT-6 interpretation guide (29), The four headache impact severity categories are little or no impact (49 or less), some impact (50-55), substantial impact (56-59), and severe impact (60-78). Range is 10-78 with higher score = more disability
Time Frame: Baseline to Immediately post-intervention
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Mindfulness Based Stress Reduction | Migraine/Stress Education
Number analyzed (Participants) | 45 | 44
score on a scale | -6.5 [-8.4 to -4.6] | -1.2 [-3.0 to 0.6]

14. Secondary Outcome: Change in Headache-related Quality of Life Scores From Baseline
Description: Change in headache-related quality of life from baseline (Migraine Specific Quality of Life, v2.1)
  The Migraine Specific Quality of Life (MSQoL) is a patient-reported outcome measure (PRO or PROM) which assesses the quality of life of migraineurs. It is a 25-item questionnaire which is filled out by the patient and is used to determine how the patient's life has been affected by their migraines - larger scores reflecting greater impact - scores ≤ 49 represent little or no impact, scores between 50 and 55 represent some impact, scores between 56 and 59 represent substantial impact, and scores ≥ 60 indicate severe impact
Time Frame: Baseline to Immediately post-intervention
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Mindfulness Based Stress Reduction | Migraine/Stress Education
Number analyzed (Participants) | 45 | 44
score on a scale | 33.6 [30.5 to 36.6] | 38.6 [35.6 to 41.6]

15. Secondary Outcome: Change in Mindfulness Scores From Baseline
Description: Change in mindfulness from baseline (Five-Facet Mindfulness Scale) - measures the trait-like tendency to be mindful in daily life. It is comprised of the following five related facets: observing, describing, acting with awareness, nonjudging, and nonreactivity - The 39 items of the Five Facet Mindfulness Questionnaire (FFMQ) are rated on a 5-point Likert scale, ranging from 1 (never or very rarely true) to 5 (very often or always true).
  * Higher scores reflect higher mindfulness scores
  * Range 39-195
  * Subscales are summed for the total score
Time Frame: Baseline to Immediately post-intervention
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Mindfulness Based Stress Reduction | Migraine/Stress Education
Number analyzed (Participants) | 45 | 44
score on a scale | 4.1 [-0.3 to 8.5] | 0.4 [-3.8 to 4.6]

16. Secondary Outcome: Change in Emotion Regulation Scores From Baseline to 12 Weeks
Description: Change in emotion regulation from baseline (Difficulty Emotion Regulation Scale), Higher scores suggest greater problems with emotion regulation - The total score ranges from 16-80 with higher scores indicating more difficulties with emotion regulation
Time Frame: Baseline to week 12
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Mindfulness Based Stress Reduction | Migraine/Stress Education
Number analyzed (Participants) | 45 | 44
score on a scale | -3.4 [-7.42 to 0.57] | 0.46 [-3.45 to 4.37]

17. Secondary Outcome: Change in Pain Catastrophizing From Baseline to 12 Weeks
Description: Change in pain catastrophizing from baseline (Pain Catastrophizing Scale)
  Patients are asked to rate the degree to which they have any of the thoughts described in the questionnaire using a 5-point Likert scale ranging from 0 (never) to 4 (always). The total score is the sum of the scores for the individual items, and ranges from 0 to 52 - higher scores relating to more pain
Time Frame: Baseline to Immediately post-intervention (12 weeks)
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Mindfulness Based Stress Reduction | Migraine/Stress Education
Number analyzed (Participants) | 45 | 44
score on a scale | -6.4 [-8.9 to -3.9] | -0.7 [-3.2 to 1.7]

18. Secondary Outcome: Change in Pain Acceptance From Baseline to 12 Weeks
Description: Change in pain acceptance from baseline (Chronic Pain Acceptance Questionnaire), higher scores reflect higher levels of pain acceptance; total range 0-156.
Time Frame: Baseline and week 12
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Mindfulness Based Stress Reduction | Migraine/Stress Education
Number analyzed (Participants) | 45 | 44
score on a scale | 5.36 [2.44 to 8.28] | 1.89 [-0.94 to 4.72]

19. Secondary Outcome: Change in Perceived Stress From Baseline to 12 Weeks
Description: Change in perceived stress from baseline (Perceived Stress Scale); Score Range: 0-40 with lower scores reflecting lower perceived stress. Ranges: 0-13 Low Stress; 14-26 Moderate Stress; 27-40 High perceived stress.
Time Frame: Baseline and week 12
Population: as for outcome 5
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Mindfulness Based Stress Reduction | Migraine/Stress Education
Number analyzed (Participants) | 45 | 44
score on a scale | -2.65 [-4.41 to -0.895] | -1.78 [-3.48 to -0.0845]

20. Secondary Outcome: Change in Depression Scores From Baseline
Description: Change in depression from baseline (Patient health-related Questionnaire-depression module, PHQ-9)
  Scores less than 5 almost always signified the absence of a depressive disorder; scores of 5 to 9 predominantly represented patients with either no depression or subthreshold (i.e., other) depression; scores of 10 to 14 represented a spectrum of patients; and scores of 15 or greater usually indicated major depression - The Patient Health Questionnaire-9 (PHQ-9) total score ranges from 0 to 27 (scores of 5-9 are classified as mild depression; 10-14 as moderate depression; 15-19 as moderately severe depression; ≥ 20 as severe depression)
Time Frame: Baseline to Immediately post-intervention
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Mindfulness Based Stress Reduction | Migraine/Stress Education
Number analyzed (Participants) | 45 | 44
score on a scale | -1.0 [-2.0 to -0.02] | 0.6 [-0.4 to 1.6]

21. Secondary Outcome: Change in Anxiety Scores From Baseline
Description: Change in anxiety from baseline (Generalized Anxiety Disorder (GAD-7). Higher Scores suggest a greater level of anxiety.
  Score 0-4: Minimal Anxiety. Score 5-9: Mild Anxiety. Score 10-14: Moderate Anxiety. Score greater than 15: Severe Anxiety - GAD-7 score of 0-4 (none), 5-9 (mild), 10-14 (moderate), and 15-21 (severe)
Time Frame: Baseline to Immediately post-intervention
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Mindfulness Based Stress Reduction | Migraine/Stress Education
Number analyzed (Participants) | 45 | 44
score on a scale | -1.6 [-2.6 to -0.5] | -0.2 [-1.2 to 0.8]

22. Secondary Outcome: Change in Self-efficacy Scores From Baseline
Description: Change in self-efficacy from baseline (Headache Management Self-Efficacy scale). Higher scores reflect more self-efficacy.
  The Headache Self-Efficacy Scale is a 51 item scale designed specifically for recurrent headache sufferers. It assesses individuals' belief that they are able to do the things necessary to prevent a moderately painful headache when confronted with personally relevant headache precipitants - The scale has a range of scores from 0-90. A higher number on the score represents a higher self-efficacy for exercise
Time Frame: Baseline to Immediately post-intervention
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Mindfulness Based Stress Reduction | Migraine/Stress Education
Number analyzed (Participants) | 45 | 44
score on a scale | 15.6 [9.2 to 22.1] | 6.8 [0.6 to 13.0]

23. Secondary Outcome: Change in Hope Scores From Baseline to 12 Weeks
Description: Change in hope from baseline (Herth Hope Index); Higher scores suggest higher levels of "Hope."
  Herth Hope Scale (HHS) is a measure that attempts to capture the multidimensional aspects of hope. This is a 4-point summated rating scale.
  Each item in the 30-item instrument is scored on a scale from 0 to 3, a score of 3 indicates that the item often applies and a score of 0 indicates that the statement never applies to the respondent. Summative scores can range from 0 to 90; higher scores denote greater hope. In terms of item order, no two consecutive items are from the same subscale.
Time Frame: Baseline and week 12
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Mindfulness Based Stress Reduction | Migraine/Stress Education
Number analyzed (Participants) | 45 | 44
score on a scale | 0.165 [-0.94 to 1.27] | -0.046 [-1.131 to 1.039]

24. Secondary Outcome: Change in Optimism From Baseline to 12 Weeks
Description: Change in optimism from baseline (Life Orientation Test-revised); Higher scores indicate greater levels of optimism.
  The Life Orientation Test (LOT) was developed to measure individual differences in optimism versus pessimism. Response options: 5-point Likert scale ranging from 0, "Strongly disagree" to 4, "Strongly agree". Total score: Items are summed, yielding a range from 0 to 32.
Time Frame: Baseline to week 12
Population: as for outcome 5
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Mindfulness Based Stress Reduction | Migraine/Stress Education
Number analyzed (Participants) | 45 | 44
score on a scale | -0.771 [-1.61 to 0.067] | -0.171 [-0.993 to 0.65]

25. Secondary Outcome: Change in Sleep From Baseline - (NIH Promis Sleep Disturbance) to Week 12
Description: Change in sleep from baseline measured with by NIH Promis Sleep Disturbance; Higher scores indicate greater severity of sleep disturbance; Range from 8-40.
Time Frame: Baseline and week 12
Population: as for outcome 5
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Mindfulness Based Stress Reduction | Migraine/Stress Education
Number analyzed (Participants) | 45 | 44
score on a scale | -1.68 [-3.29 to -0.079] | 0.9784 [-0.601 to 2.558]

26. Secondary Outcome: Change in Sleep From Baseline - (NIH Promis Sleep Disturbance) to 12 Weeks
Description: as for outcome 25
Time Frame: Baseline and week 12
Population: Data were not collected
Arm/Group | Mindfulness Based Stress Reduction | Migraine/Stress Education
Number analyzed (Participants) | 0 | 0

27. Secondary Outcome: Change in Global Health From Baseline to 12 Weeks
Description: Change in global health from baseline (NIH Promis Global Health-1st question); Range 0-5, 5 highest.
Time Frame: Baseline and week 12
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Mindfulness Based Stress Reduction | Migraine/Stress Education
Number analyzed (Participants) | 45 | 44
score on a scale | 3.48 [3.23 to 3.74] | 3.23 [2.98 to 3.48]

28. Secondary Outcome: Change in Social Connectedness From Baseline to 12 Weeks
Description: Change in social connectedness from baseline (Social Connectedness Scale-revised); Higher scores reflect a higher level of social connection.
  It is on a likert scale with 1 being strongly disagree to 6 being strongly agree.
Time Frame: Baseline to week 12
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Mindfulness Based Stress Reduction | Migraine/Stress Education
Number analyzed (Participants) | 45 | 44
score on a scale | -1.00 [-3.57 to 1.56] | -.447 [-2.97 to 2.08]

29. Secondary Outcome: Change in Flourishing From Baseline to 12 Weeks
Description: Change in flourishing from baseline (Flourishing scale); Higher scores represents a person with many psychological resources and strength; Range from 8-56.
Time Frame: Baseline and week 12
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Mindfulness Based Stress Reduction | Migraine/Stress Education
Number analyzed (Participants) | 45 | 44
score on a scale | 1.07 [-0.710 to 2.85] | -0.10 [-1.85 to 1.65]

30. Secondary Outcome: Change in Resilience Scores From Baseline to 12 Weeks
Description: Change in resilience from baseline (Brief Resilience scale); higher scores indicate greater levels of resilience; scores range from 6-30
Time Frame: Baseline to week 12
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Mindfulness Based Stress Reduction | Migraine/Stress Education
Number analyzed (Participants) | 45 | 44
score on a scale | 0.238 [-0.793 to 1.269] | -0.486 [-1.497 to 0.525]

31. Secondary Outcome: Change in Allodynia From Baseline to 12 Weeks
Description: Change in allodynia from baseline (Allodynia Symptom Checklist), score range 0-24, 0-2 none; 3-5 mild; 6-8 moderate; 9+ severe
  Cutaneous allodynia (CA) scale defining no CA (scores 0-2), mild CA (3-5), moderate CA (6-8), and severe CA (≥9).
Time Frame: Baseline to week 12
Population: Data were not collected
Arm/Group | Mindfulness Based Stress Reduction | Migraine/Stress Education
Number analyzed (Participants) | 0 | 0

32. Secondary Outcome: Change in Number of Migraine Days From Baseline
Description: as for outcome 1
Time Frame: Baseline to 6 months post-intervention
Measure: Mean (95% Confidence Interval); unit: change in the number of days
Arm/Group | Mindfulness Based Stress Reduction | Migraine/Stress Education
Number analyzed (Participants) | 45 | 44
change in the number of days | -2.2 [-3.2 to -1.2] | -2.7 [-3.8 to -1.7]

33. Secondary Outcome: Change in Number of Headache Days From Baseline
Description: Change in frequency of any day with a headache tracked with headache logs
Time Frame: Baseline to 3 Months post-intervention
Measure: Mean (95% Confidence Interval); unit: change in Number of days
Arm/Group | Mindfulness Based Stress Reduction | Migraine/Stress Education
Number analyzed (Participants) | 45 | 44
change in Number of days | -3.18 [-4.3 to -2.0] | -3.7 [-4.8 to -2.5]

34. Secondary Outcome: Change in Number of Headache Days From Baseline
Description: Change in frequency of any day with a headache tracked with headache logs
Time Frame: Baseline to 6 Months post-intervention
Measure: Mean (95% Confidence Interval); unit: change in Number of days
Arm/Group | Mindfulness Based Stress Reduction | Migraine/Stress Education
Number analyzed (Participants) | 45 | 44
change in Number of days | -3.2 [-4.4 to -1.9] | -4.1 [-5.4 to -2.8]

35. Secondary Outcome: Change in Headache Duration From Baseline to 24 Weeks
Description: Modeled change in headache duration from baseline 4 weeks to weeks 20-24 by calculating the duration (in hours) of each headache attack
Time Frame: Baseline to 3 Months post-intervention (24 weeks)
Population: Data were not collected
Arm/Group | Mindfulness Based Stress Reduction | Migraine/Stress Education
Number analyzed (Participants) | 0 | 0

36. Secondary Outcome: Change in Headache Duration From Baseline to 36 Weeks
Description: Modeled change in headache duration from baseline 4 weeks to weeks 32-36 by calculating the duration (in hours) of each headache attack
Time Frame: Baseline to 6 Months post-intervention (36 weeks)
Population: Data were not collected
Arm/Group | Mindfulness Based Stress Reduction | Migraine/Stress Education
Number analyzed (Participants) | 0 | 0

37. Secondary Outcome: Change in Headache Severity-pain Intensity From Baseline to 24 Weeks
Description: change in headache severity-pain intensity from baseline 4 weeks to weeks 20-24 weeks. For each headache attack, participants rated the pain intensity on a 0-10 scale (0, no pain sensation, 10 most intense pain sensation imaginable). We calculated the pain intensity of each headache attack and used a multivariable linear mixed model framework controlling for baseline value of the outcome of interest, treatment group, cohort, and within participant variation via random effects, with significance based on the treatment group effect and phase interaction at .05 significance level.
Time Frame: Baseline and 24 weeks
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Mindfulness Based Stress Reduction | Migraine/Stress Education
Number analyzed (Participants) | 45 | 44
score on a scale | 0.111 [-0.238 to 0.460] | -0.1666 [-0.509 to 0.178]

38. Secondary Outcome: Change in Headache Severity-pain Intensity From Baseline to 36 Weeks
Description: change in headache severity-pain intensity from baseline 4 weeks to weeks 32-36. For each headache attack, participants rated the pain intensity on a 0-10 scale (0, no pain sensation, 10 most intense pain sensation imaginable). We calculated the pain intensity of each headache attack and used a multivariable linear mixed model framework controlling for baseline value of the outcome of interest, treatment group, cohort, and within participant variation via random effects, with significance based on the treatment group effect and phase interaction at .05 significance level.
Time Frame: Baseline and 36 weeks
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Mindfulness Based Stress Reduction | Migraine/Stress Education
Number analyzed (Participants) | 45 | 44
score on a scale | 0.1049 [-0.374 to 0.584] | 0.047 [-0.473 to 0.567]

39. Secondary Outcome: Change in Headache Severity-pain Unpleasantness From Baseline to 24 Weeks
Description: Change in headache severity on 0-10 scale (0, "not at all unpleasant" to 10, "most unpleasant imaginable") in pain unpleasantness from baseline 4 weeks to weeks 20-24 (tracked with headache logs).
Time Frame: Baseline and 24 weeks
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Mindfulness Based Stress Reduction | Migraine/Stress Education
Number analyzed (Participants) | 45 | 44
score on a scale | -0.107 [-0.499 to 0.285] | -0.046 [-0.432 to 0.340]

40. Secondary Outcome: Change in Headache Severity-pain Unpleasantness From Baseline to Week 36
Description: Change in headache severity on 0-10 scale (0, "not at all unpleasant" to 10, "most unpleasant imaginable") in pain unpleasantness from baseline 4 weeks to weeks 32-36 (tracked with headache logs).
Time Frame: Baseline and week 36
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Mindfulness Based Stress Reduction | Migraine/Stress Education
Number analyzed (Participants) | 45 | 44
score on a scale | -0.0811 [-0.573 to 0.411] | 0.0977 [-0.437 to 0.632]

ADVERSE EVENTS:
Time Frame: 36 weeks
Description: Adverse events were systematically queried and tracked at each study visit.
Arm/Group | Mindfulness Based Stress Reduction | Migraine/Stress Education
All-Cause Mortality (participants affected / at risk) | 0/45 | 0/44
Serious Adverse Events (participants affected / at risk) | 0/45 | 0/44
Other Adverse Events (participants affected / at risk) | 1/45 | 0/44
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mindfulness Based Stress Reduction (N=45) | Migraine/Stress Education (N=44)
squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) — One MBSR participant developed squamous cell carcinoma, deemed unrelated to the study protocol.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-02-19): https://cdn.clinicaltrials.gov/large-docs/98/NCT02695498/Prot_SAP_001.pdf
  • Informed Consent Form (2018-09-18): https://cdn.clinicaltrials.gov/large-docs/98/NCT02695498/ICF_002.pdf